CLINICAL TRIAL: NCT01628861
Title: Point-of-Choice Prompts to Reduce Prolonged Sitting Time at Work: A Randomised Trial
Brief Title: Point-of-Choice Prompts to Reduce Prolonged Sitting Time at Work
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Principal Investigator, Philippa Dall, PhD, Research Fellow, Glasgow Caledonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 200813897
Record Dates: First submitted 2012-06-22; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Adult Office Workers
Keywords: occupation; work; sitting; sedentary behaviour; office worker; adult; education; point-of-choice prompt

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- education only (Active Comparator): A short educational talk, read from a script, regarding the health risks of prolonged sitting, stating that standing every 30 minutes could be beneficial. A short information leaflet with the same message is also provided.
  Interventions: Behavioral: education talk and leaflet
- prompt + education (Experimental): A short educational talk, read from a script, regarding the health risks of prolonged sitting, stating that standing every 30 minutes could be beneficial. A short information leaflet with the same message is also provided. Prompting software (MyRestBreak 1.0 copyright Vikram Sharma) will be installed on the work computer. A prompt with the message "stand up, take a break" is placed on the screen of the work computer for 1 minutes every 30 minutes, from the time the computer is switched on in the morning. The prompt is contained in a window 11x9 cm in the centre of the screen. The prompt cannot be removed or minimised, but work can continue in any windows visible around the prompt. The prompt is on the computer for 5 days.
  Interventions: Device: MyRestBreak 1.0; Behavioral: education talk and leaflet

INTERVENTIONS:
Device: MyRestBreak 1.0 — Prompting software (MyRestBreak 1.0 copyright Vikram Sharma) will be installed on the work computer. A prompt with the message "stand up, take a break" is placed on the screen of the work computer for 1 minutes every 30 minutes, from the time the computer is switched on in the morning. The prompt is contained in a window 11x9 cm in the centre of the screen. The prompt cannot be removed or minimised, but work can continue in any windows visible around the prompt. The prompt is on the computer for 5 days.
  Arms: prompt + education
Behavioral: education talk and leaflet — A short educational talk, read from a script, regarding the health risks of prolonged sitting, stating that standing every 30 minutes could be beneficial. A short information leaflet stating with the same message is also provided.

SUMMARY:
The purpose of this study is to determine whether an on-screen prompt put on the work computer every 30 minutes is effective in getting office workers to reduce prolonged periods of sitting at work.

DETAILED DESCRIPTION:
Prolonged bouts of uninterrupted time spent sitting is associated with indicators of poor health, independent of how physically active a person is. Many occupations are now sedentary, and are characterised by long periods spent sitting at a desk. Brief education on the benefits of standing regularly and breaking up prolonged sitting will be provided to participants, working at a Scottish University. One intervention group will additionally have software installed on their work computer which placed a prompt window in the centre of their screen for 1 minute every 30 minutes. The prompt will remind participants to stand-up and take a break, and the window cannot be removed or minimised.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Glasgow Caledonian University
* Aged between 18 and 65 years
* Self-reported desk-based occupation
* Informed written consent provided
* Ability to stand unassisted

Exclusion Criteria:

* Any musculoskeletal condition which limits ability to stand regularly

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
duration of prolonged sitting | 5 days
  total time spent sitting in continuous uninterrupted prolonged (>30minutes) sitting events at work

SECONDARY OUTCOMES:
total sitting duration | 5 days
  total time spent sitting while at work
number of sitting events | 5 days
  total number of uninterrupted sitting events (of any duration) during work
step count | 5 days
  total number of steps taken while at work
break duration | 5 days
  the duration of breaks between sitting events
walking time | 5 days
  total time spent walking at work
standing time | 5 days
  total time spent standing while at work
number of prolonged sitting events | 5 days
  the number of continuous uninterrupted prolonged (>30minutes) sitting events during work

CONTACTS AND LOCATIONS:
Overall Officials: Philippa M Dall, PhD, Principal Investigator — Glasgow Caledonian University
Locations (1):
- School of Health & Life Sceinces, Glasgow Caledonian University, Glasgow, Lanarkshire, United Kingdom

REFERENCES:
- [Derived] Evans RE, Fawole HO, Sheriff SA, Dall PM, Grant PM, Ryan CG. Point-of-choice prompts to reduce sitting time at work: a randomized trial. Am J Prev Med. 2012 Sep;43(3):293-7. doi: 10.1016/j.amepre.2012.05.010. PMID 22898122